CLINICAL TRIAL: NCT02278393
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL STUDY TO EVALUATE THE SAFETY OF EXCESSIVE CONSUMPTION OF PLANT STEROL-ENRICHED FERMENTED DAIRY PRODUCT OVER A 4-WEEK PERIOD IN JAPANESE HEALTHY ADULTS
Brief Title: A Clinical Study for Evaluating the Safety of a Plant Sterol-enriched Fermented Dairy Product in Japanese Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Japan (Industry)
Responsible Party: Sponsor
Organization: Danone Global Research & Innovation Center (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: NU360
Record Dates: First submitted 2014-10-16; First posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
Keywords: Japanese healthy volunteers; High LDL-C; dairy drinks; phytosterols
MeSH Terms: interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Fermented Dairy Product with Phytosterols (test) (Active Comparator): one arm active = 3 bottles of test product/day with 1,6g of phytosterols each
  Interventions: Other: 1-Fermented Dairy Product with Phytosterols (test)
- 2-Fermented dairy Product with No Phytosterols (control) (Placebo Comparator): one arm control product= 3 bottles test productl/day with no Phytosterols
  Interventions: Other: 2-Fermented dairy Product with No Phytosterols (control)

INTERVENTIONS:
Other: 1-Fermented Dairy Product with Phytosterols (test) — 1- 3 bottles of test product/day
  Arms: 1-Fermented Dairy Product with Phytosterols (test)
Other: 2-Fermented dairy Product with No Phytosterols (control) — 2-3 bottles of control product/day
  Arms: 2-Fermented dairy Product with No Phytosterols (control)

SUMMARY:
Investigate the safety of excessive consumption of plant sterol-enriched fermented dairy product over a 4-week period in Japanese healthy adults

ELIGIBILITY:
Inclusion Criteria:

* To be checked at the inclusion visit (V1) :
* II 01: Male/female subject, aged from 20 to 55 years (bounds included).
* II 02: Subject with body mass index (BMI) between 18.5 kg/m2 (bound included) and 30 kg/m2 (bound excluded).
* II 03: Subject with LDL-cholesterol plasma level under 140 mg/dL (3.6 mmol/L) (bound excluded).
* II 04: Subject with triglycerides under 200 mg/dL (2.3 mmol/L) (bound included).
* II 05: Non hypertensive subject defined with Systolic Blood Pressure (SBP) <140mmHg and Diastolic Blood Pressure (DBP) <90 mmHg.
* II 06: Subject agreeing not to consume any supplements/excessive plant sterols and plant stanols in any form during the study period.
* II 07: If of childbearing potential, female subject must be using or complying with one of the following medically approved methods of contraception such as, but not exclusively:
* Oral birth control pills (at least 1 full monthly cycle prior to study product administration);
* Intra-uterine device (IUD);
* Double barrier methods (such as condoms and spermicide); OR female subject must be postmenopausal for at least 12 months prior to trial entry or surgically sterile (i.e. hysterectomy, bilateral oophorectomy or bilateral tubal ligation).
* II 08: Subject covered by social security or covered by similar system.
* II 09: Subject, upon briefing of the content of the present study, fully understanding and agreeing to its objective; and being able to personally sign a written informed consent.
* II 10: Subject having given written (dated and signed) inform consent to take part in the study.
* II 11: Asian subjects originating from Japan
* II12: Subject who is able to communicate well with the investigator and to comply with the requirements of the entire study.
* II13: Subject having a fridge at home for study products storage with sufficient capacity.

To be checked at the randomization visit (V2):

- RI 01: Subject having followed the dietary recommendations over the wash-out period.

Exclusion Criteria:

* To be checked at the inclusion visit (V1):
* IE 01: Subject having experienced any cardiovascular event (cardiac infarction, angina attack, surgical or endoscopic coronary angioplasty, stroke, arterial disease, etc.).
* IE 02: Subject suffering from any serious or chronic liver, renal, cardiovascular, respiratory, endocrine or metabolic disorders.
* IE 03: Subject with gastro-intestinal disorders (such as diarrhoea, constipation, irritable bowel syndrome) or using laxatives.
* IE 04: Subject with diabetes Type I and Type II or Fasting Blood Sugar test (FBS) > 125 mg/dL at screening visit.
* IE 05: Subject with active liver disease or hepatic dysfunction as defined by elevations in liver enzymes: [alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT) > 3X the upper limit of normal (ULN).
* IE 06: Subject with unexplained serum creatine phosphokinase (CPK) > 2X the upper limit of normal (ULN). Subject with a reason for CPK elevation may continue in inclusion process and have the measurement repeated prior to randomization; a repeat CPK > 2X ULN is exclusionary.
* IE 07: Subject with weight change (variation > 5%) within 6 months at least prior to inclusion.
* IE 08: Subject taking any hypocholesterolemic drugs or products (statins, ezetimibe, sequesterants, niacin, nicotinates, probucol, omega-3 fatty acids (EPA-DHA, ALA…), and fibrates).
* IE 09: Subjects having stopped their hypocholesterolemic drugs or products for less than 3 months
* IE 10: Subject with known lactose intolerance.
* IE 11: Subject with known allergy or hypersensitivity to plant sterols and to any component of the study product (milk protein for example).
* IE 12: Subjects having sitosterolemia.
* IE 13: Subject who had any surgery or intervention requiring a general anaesthesia in the preceding 4 weeks, or who plans to have one during the course of the study.
* IE 14: Subject receiving (currently or in the 4 last weeks) systemic treatment or topical treatment likely to interfere with evaluation of the study parameters.
* IE 15: Subject involved in any other clinical study within the preceding month or in the exclusion period after another clinical study.
* IE 16 Subject having blood sample of 200 mL or more taken (e.g., donated blood) within 1 month, or 400 mL or more within 3 months before the start of the present study.
* IE 17: Subject with heavy alcohol intake (> 60 g/day).
* IE 18: Subject taking any treatment for anorexia, weight loss, or any form of treatment likely to interfere with metabolism or dietary habits (e.g. hypolipemic, hypoglycaemic treatments).
* IE 19: For female subject: pregnant woman or woman planning to become pregnant during the study; breast-feeding woman.
* IE 20: For female subject: subject likely to change her contraceptive method or hormone replacement therapy during the study.
* IE 21: Subject in a situation, which in the investigator's opinion could interfere with optimal participation in the present study (e.g. -products consumer) or could constitute a special risk for the subject.
* IE 22: Subject who is susceptible to not comply with dietary qualitative restriction during the study period.
* IE 23 Vulnerable subjects defined as individuals whose willingness to volunteer in the clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. Examples are members of a group with a hierarchical structure, such as medical, pharmacy, dental and nursing students, subordinate hospital and laboratory personnel, employees of the pharmaceutical industry, members of the armed forces, and persons kept in detention.
* IE 24: Subject expected to be living in the same home as a current participating subject and to concomitantly receive some study products.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From baseline to 6 weeks (4-week consumption + 2-week follow-up periods)
  Number of subjects with at least one adverse event by study group

SECONDARY OUTCOMES:
Adverse Events | From baseline to 6 weeks (4-week consumption + 2-week follow-up periods)
  Number of adverse events by study group
Vital signs | From baseline to 6 weeks (4-week consumption + 2-week follow-up periods)
  Descriptive statistics for systolic and diastolic blood pressure, heart rate and BMI
Vital signs | From baseline to 6 weeks (4-week consumption + 2-week follow-up periods)
  To assess the change for systolic and diastolic blood pressure, heart rate and BMI
Laboratory measurements | From baseline to 6 weeks (4-week consumption + 2-week follow-up periods)
  Descriptive statistics for Haematology parameters, liver/kidney/muscle function parameters, carbohydrate metabolism parameters, lipids, minerals, proteins and electrolytes
Laboratory measurements | From baseline to 6 weeks (4-week consumption + 2-week follow-up periods)
  To assess the change for Haematology parameters, liver/kidney/muscle function parameters, carbohydrate metabolism parameters, lipids, minerals, proteins and electrolytes

CONTACTS AND LOCATIONS:
Overall Officials: Christine MRINI, MD, PHD, Study Director — Danone Research Life Sciences
Locations (1):
- Yaesu Sakura-dori Clinic, Tokyo, Japan